CLINICAL TRIAL: NCT05011916
Title: An Exploratory Clinical Study on the Safety and Efficacy of KDR2-2 Suspension Eye Drops in the Treatment of Corneal Neovascularization
Brief Title: The Safety and Efficacy of KDR2-2 Suspension Eye Drops in the Treatment of Corneal Neovascularization
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021KYPJ139
Record Dates: First submitted 2021-08-07; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization

STUDY DESIGN:
Intervention Model Description: 4
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Patients in the control group received 0.1% fluorometholone eye drops (0.1% fluorometholone + 0.05% tacrolimus eye drops for patients after corneal transplantation). The patients applied 0.1% fluorometholone eye drops 4 times daily for 10 weeks. Patients were instructed to continue with their usual ophthalmic medication regimens, such as topical antibacterial and antiviral drugs.
- Low-concentration group (Experimental): Patients in the low-concentration group applied 4mg/ml KDR2-2 suspension eye drops 4 times daily for 6 weeks. The rest of the medication regimen is the same as the control group.
  Interventions: Drug: KDR2-2 suspension eye drops
- Medium-concentration group (Experimental): Patients in the medium-concentration group applied 4mg/ml KDR2-2 suspension eye drops 4 times daily for 6 weeks. The rest of the medication regimen is the same as the control group.
  Interventions: Drug: KDR2-2 suspension eye drops
- High-concentration group (Experimental): Patients in the High-concentration group applied 4mg/ml KDR2-2 suspension eye drops 4 times daily for 6 weeks. The rest of the medication regimen is the same as the control group.
  Interventions: Drug: KDR2-2 suspension eye drops

INTERVENTIONS:
Drug: KDR2-2 suspension eye drops — All patients were instructed to instill one drop four times per day in the study eye for 6 weeks.
  Arms: High-concentration group; Low-concentration group; Medium-concentration group

SUMMARY:
KDR2-2, as a tyrosine kinase inhibitor, has a strong inhibitory effect on VEGFR2 and a moderate inhibitory effect on PDGFR-β. It can be used for the treatment of corneal neovascularization. The main purpose of this study is to explore the efficacy and safety of KDR2-2 suspension eye drops in the treatment of corneal neovascularization. This study is a single-center, prospective, randomized controlled clinical study. A total of 60 patients with corneal neovascularization were enrolled in this study, and they were randomly divided into 4 groups, including the control group, the KDR2-2 low-concentration (4mg/ml) group, the medium-concentration (10mg/ml) group, and the high-concentration (20mg/ml) group, with 15 subjects in each group. The control group applied 0.1% fluorometholone eye drops, and the test groups applied KDR2-2 suspension eye drops with 0.1% fluorometholone eye drops. Patients applied KDR2-2 eye drops four times daily for 6 weeks and were followed up to 10 weeks. The follow-up time points were baseline, 1 week, 2 weeks, 4 weeks, 6 weeks after medication, and 4 weeks after drug withdrawal. Relevant ophthalmological examinations (including visual acuity, intraocular pressure, slit lamp microscopy, central corneal thickness measurement, corneal fluorescein staining assessment, corneal sensitivity measurement, corneal confocal microscope examination, and anterior segment and fundus photography) are performed at each time. And the ocular tolerability score and adverse events of each patient were recorded. By comparative analysis, the efficacy and safety of KDR2-2 eye drops in the treatment of corneal neovascularization were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily participate in the trial, sign the informed consent form, and follow up according to the time specified by the trial;
2. 18~75 years old, without gender limit;
3. Superficial or deep corneal progressive neovascularization induced by trauma, chemical burns, corneal transplantation and inflammation: the growth of corneal new vessels≥ 2 mm from the limbus within 1 week to 2 months.

Exclusion Criteria:

1. Obvious corneal epithelial defects (>1mm), or a history of persistent corneal epithelial defects in the past 3 months (>1mm, ≥14 days);
2. Anti-VEGF drugs have been injected locally in the target eye within 3 months, or anti-VEGF drugs have been used systemically within 2 months;
3. Recent eye surgery (except for keratoplasty) within 3 months, or planned eye surgery during the trial period;
4. Systemic use of glucocorticoid drugs, or intraocular or periocular injection of glucocorticoid drugs within 1 month;
5. Contact lenses use within the past 2 weeks (except bandage lenses);
6. Stable corneal neovascularization: > 6 months;
7. History of coagulation abnormalities (such as end-stage liver disease), or current anticoagulant drugs other than aspirin (such as warfarin, heparin, enoxaparin or similar anticoagulants);
8. Uncontrolled clinical problems (such as tumors, HIV infection, hepatitis C virus infection, active hepatitis B or other serious chronic infections, serious mental, neurological, cardiovascular, urinary, respiratory and other system diseases, etc.); Uncontrolled hypertension: systolic blood pressure ≥150mmHg or diastolic blood pressure ≥90mmHg; uncontrolled diabetes: A1C>7%;
9. Unwillingness/inability to take effective contraceptive measures during the trial period;
10. Female subjects have a positive blood pregnancy test;
11. Participated in a drug clinical trial within 3 months;
12. The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-08-09 (Estimated); Study Completion 2022-08-09 (Estimated)

PRIMARY OUTCOMES:
the changes of the size and extent of corneal neovascularization | Baseline, 1 week, 2 weeks, 4 weeks and 6 weeks after medication, and 4 weeks after drug withdrawal
  The efﬁcacy of KDR2-2 eye drops treatment on corneal neovascularization was evaluated by comparing corneal anterior segment photographs acquired at baseline with photographs acquired on the follow-up visits. Size and extent of CNV was investigated by four primary metrics: (1) neovascular area ratio, the ration of the area of the neovascularization to the area of the cornea, (2) vessel length (VL), the total length of the vessels projected into the cornea, (3) vessel caliber, the mean diameter of the corneal vessels, and (4) Corneal neovascularization progression/stabilization/regression rate

SECONDARY OUTCOMES:
the changes of visual acuity | Baseline, 1 week, 2 weeks, 4 weeks and 6 weeks after medication, and 4 weeks after drug withdrawal
  The uncorrected visual acuity and best corrected visual acuity were assessed through ETDRs chart at baseline and all the follow-up visits. The alterations in visual acuity were evaluated in all patients.
the changes of intraocular pressure | Baseline, 1 week, 2 weeks, 4 weeks and 6 weeks after medication, and 4 weeks after drug withdrawal
  The intraocular pressure of the patients was assessed by iCARE at baseline and all the follow-up visits. The alterations of intraocular pressure were evaluated.
the changes of central corneal thickness | Baseline, 1 week, 2 weeks, 4 weeks and 6 weeks after medication, and 4 weeks after drug withdrawal
  The central corneal thickness was assessed by anterior segment OCT at baseline and all the follow-up visits. The alterations in central corneal thickness were evaluated.
the changes of conjunctival hyperemia score | Baseline, 1 week, 2 weeks, 4 weeks and 6 weeks after medication, and 4 weeks after drug withdrawal
  The conjunctival hyperemia score was assessed by severity from 0 (no signs of conjunctival hyperemia) to 3 (serious conjunctival hyperemia) by the clinician at baseline and all the follow-up visits.The changes of conjunctival hyperemia score were evaluated.
the changes of corneal fluorescein staining score | Baseline, 1 week, 2 weeks, 4 weeks and 6 weeks after medication, and 4 weeks after drug withdrawal
  The corneal fluorescein staining score was assessed by NEI grading system by the clinician at baseline and all the follow-up visits.The NEI grading system divides the cornea into 5 zones: central, superior, temporal, nasal, and inferior. For each zone, the amount of corneal ﬂuorescein staining is graded on a scale of 0 to 3: 0=normal or negative slit-lamp ﬁndings; 1=milder superfacial stippling; 2=moderate or punctate staining, including superfacial abrasion of the cornea; and 3=severe abrasion or corneal erosion, deep corneal abrasion, or recurrent erosion. The alterations in corneal fluorescein staining score were evaluated.
the changes of corneal sensation | Baseline and 4 weeks after drug withdrawal
  The corneal sensation was assessed through Cochet-Bonnet aesthesiometer by the clinician at baseline and 4 weeks after drug withdrawal. The corneal sensation was assessed at five points on the cornea, including the central, superior, temporal, nasal, and inferior points.
the morphological changes of corneal subepithelial nerve | Baseline and 4 weeks after drug withdrawal
  In vivo confocal laser scanning microscopy was performed by the clinician at baseline and 4 weeks after drug withdrawal. The density and length of the corneal subepithelial nerve were analysed.
the changes of ocular tolerability score | 1 week, 2 weeks, 4 weeks and 6 weeks after medication
  Ocular tolerability score (including ocular tolerability, burning sensation, pain, itching and blurred vision) was assessed by severity from 0 (absent) to 3 (severe) by questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan Opthalmic Center, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou